CLINICAL TRIAL: NCT06001333
Title: Efficacy and Safety of Fecal Microbiota Transplantation for the Decolonization of Multidrug-Resistant Organisms in the Intestinal Tract: An Unblinded Randomized Controlled Trial
Brief Title: Efficacy and Safety of FMT for the Decolonization of MDROs in the Intestinal Tract
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chuncheon Sacred Heart Hospital (Other)
Collaborators: Severance Hospital (Other); National Institute of Health, Korea (Other Government)
Responsible Party: Principal Investigator, Seung Soon Lee, Associate Professor, Chuncheon Sacred Heart Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-06-007
Record Dates: First submitted 2023-08-14; First posted 2023-08-21 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Carbapenem-Resistant Enterobacteriaceae; Vancomycin (Glycopeptide) Resistant Enterococcus (VRE)
Keywords: Carbapenem-Resistant Enterobacteriaceae; Vancomycin-Resistant Enterococci; Fecal Microbiota Transplantation; Gastrointestinal Microbiome
MeSH Terms: interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- FMT group (Experimental): fecal microbiota transplantation using frozen or capsulized stool
  Interventions: Procedure: fecal microbiota transplantation
- non-FMT group (No Intervention): Simple observation without intervention

INTERVENTIONS:
Procedure: fecal microbiota transplantation — Fecal microbiota transplantation will be conducted on patients using donor stool (frozen or capsulized stool) from a stool bank.
  Arms: FMT group

SUMMARY:
The goal of this unblinded randomized controlled trial is to evaluate the efficacy and safety of fecal microbiota transplantation for the decolonization of carbapenemase-producing carbapenem-resistant Enterobacteriaceae (CP-CRE) or vancomycin-resistant Enterococci (VRE) in the intestinal tract. The study is planned to be conducted to test the superiority hypothesis that the decolonization success rate in the FMT group is higher compared to the non-FMT group. Outcome analysis will be conducted through intention-to-treat analysis, modified intention-to-treat analysis, and per-protocol analysis.

The main questions it aims to answer are:

* primary endpoint: Rate of Decolonization of Multidrug-Resistant Organisms (CP-CRE or VRE) at 1 Month After Fecal Microbiota Transplantation (FMT).
* secondary endpoint: Rates of Multidrug-Resistant Organism decolonization at 3 months, 6 months, and 1 year after FMT / Post-FMT Multidrug-Resistant Organism Recolonization Rate and Infection Rate.

Patients colonized with multidrug-resistant organisms in the gastrointestinal tract are divided into two groups through obtaining written consent from the patients and random allocation: the Fecal Microbiota Transplantation group (FMT group), which receives FMT, and the control group (non-FMT group), which is observed without FMT. The decolonization status of multidrug-resistant organisms will be monitored every 3-7 days after FMT until three consecutive negative results.

DETAILED DESCRIPTION:
The study is planned to be conducted at Chuncheon Sacred Heart Hospital and Severance Hospital, using randomization with equal allocation to allocate patients into FMT (Fecal Microbiota Transplantation) and non-FMT groups. The study parameters are set with an alpha error of 0.05 and beta error of 0.2. Considering the findings from previous research, a delta value (effect size) was determined for sample size calculation. Based on this calculated sample size, for CP-CRE, 80 patients will be recruited in the FMT group compared to 68 patients in the non-FMT group. For VRE, 48 patients will be recruited in the FMT group compared to 44 patients in the non-FMT group.

Patients who have provided written consent for participation in the study will be required to maintain fasting starting from the evening before the procedure, after discontinuing broad-spectrum antibiotics for a minimum of 3-7 days. Subsequently, a bowel preparation will be carried out twice - the evening before and the morning of the procedure. Once the bowel preparation is complete, 1 hour before the procedure, patients will receive loperamide to reduce bowel movements and then proceed to the endoscopy suite.

Fecal microbiota transplantation (FMT) will be carried out with the acquired frozen donor stool, which will be thawed for 2 hours at room temperature following purchase and delivery from a stool bank, under the consent and supervision of the patient or guardian. Frozen stool from carefully screened donors who have passed the rigorous screening of both Stage 1 clinical assessment and Stage 2 laboratory tests (including evaluation for antibiotic resistance organisms) will be supplied from a stool bank of Microbiotix inc.

The FMT procedure will be conducted in collaboration with the research team in the Division of Gastroenterology. During the procedure, no tissue biopsy or excessive endoscope insertion will be performed. The FMT involves the simple infusion of thawed donor stool into the terminal ileum under colonoscopy, which takes approximately 5-10 minutes. The procedure carries minimal risk of bleeding, perforation, or aspiration. In most cases, it will be performed under sedation with a colonoscopy. If smooth insertion of the colonoscope or proper visualization of the colon is hindered, or if colonic preparation is not successful, Esophagogastroduodenoscopy (EGD) will be performed with sedation, and thawed donor stool will be infused into the third portion of the duodenum. This procedure also poses minimal risk of regurgitation or aspiration due to its anatomical and physiological characteristics. After the procedure, the lower extremities will be elevated by about 30 degrees to prevent the transplanted stool from exiting. A one-day fasting period will be maintained after the procedure to facilitate successful engraftment of the transplanted stool, followed by the gradual resumption of a regular diet. Following FMT, repeated rectal swab cultures will be conducted to confirm three consecutive negative results for CP-CRE or VRE at 3-7 day intervals.

In cases where encapsulated fecal material is used for FMT, it will be ingested along with high-acid cranberry or orange juice. The capsules are specially designed to dissolve in low-acidic environments, allowing them to reach the terminal ileum for safe administration without the need for bowel preparation. On the first day, 15 capsules will be consumed, followed by another 15 capsules on the second day, for a total of 30 capsules. Subsequently, repeated rectal swab tests will be conducted to confirm three consecutive negative results for CP-CRE or VRE at 3-day intervals.

According to patient random allocation, fecal samples and clinical metadata will be periodically collected (prior to FMT, 1 month, 3 months, 6 months, and 12 months after FMT) from both recipients and donors. These collected samples will undergo full-length 16S rRNA sequencing and shotgun metagenomic sequencing to comprehensively analyze the gut microbiome. Through this analysis, the aim is to elucidate the intestinal microorganisms associated with decolonization outcome and their mechanisms.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals aged 20 and older.
2. Those with confirmed carbapenemase-producing Enterobacteriaceae (CPE) from a rectal swab culture within the past week (class A, B, or D CPE).
3. Those with confirmed vancomycin-resistant Enterococci (E. fecalis or E. faecium) from a rectal swab culture within the past week.
4. Individuals who have agreed to undergo Fecal Microbiota Transplantation (FMT) procedures and to provide pre- and post-procedure stool samples.
5. Individuals who have discontinued antibiotics for a period of 3 to 7 days prior to FMT procedure.

Exclusion Criteria:

1. Patients with ongoing or anticipated acute treatment, including antibiotic therapy.
2. Individuals with severe immunodeficiency.
3. Cases where there is a risk due to upper gastrointestinal endoscopy or colonoscopy.
4. Pregnant individuals, those who could become pregnant, and breastfeeding women.
5. Cases where participation in the study is determined by the researcher not to be beneficial.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-09-18 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of Decolonization of Multidrug-Resistant Organisms at 1 Month After Fecal Microbiota Transplantation (FMT) | at 1 Month After Fecal Microbiota Transplantation (FMT)
  The decolonization rate at 1 month after FMT refers to the proportion of achieving three consecutive negative results within 1 month after the FMT procedure.

SECONDARY OUTCOMES:
rates of Multidrug-Resistant Organism decolonization at 3 months, 6 months, and 1 year after Fecal Microbiota Transplantation (FMT) | at 3 months, 6 months, and 1 year after Fecal Microbiota Transplantation (FMT)
  The decolonization rate at 1 month, 3 months, and 1 year after FMT refers to the proportion of achieving three consecutive negative results within 3 months, 6 months, and 12 months after the FMT procedure.
Post-FMT Multidrug-Resistant Organism Recolonization Rate and Infection Rate within 1 year after FMT | within 12 months after FMT
  The rates of re-colonization of decolonized multidrug-resistant organisms (CP-CRE or VRE) and clinical infection rates of MDROs within 1 year after FMT procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Seung Soon Lee, MD, PhD, Principal Investigator — Chuncheon Sacred Heart Hospital
Locations (2):
- South Korea (2):
  - Chuncheon Sacred Heart Hospital, Chuncheon, Gangwon-do
  - Severance Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No